CLINICAL TRIAL: NCT01679145
Title: Learning Mechanisms as Predictors of Treatment Outcome in Alcohol- Dependent Patients
Brief Title: Learning and Relapse Risk in Alcohol Dependence
Acronym: LeAD
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Charite University, Berlin, Germany (Other); University Hospital Carl Gustav Carus (Other)
Responsible Party: Sponsor
Other Study IDs: HE2597/141;ZI1119/31;WI709/101
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Alcohol Use Disorders
Keywords: Reward- based learning; Pavlovian-to-instrumental transfer; Functional imaging; Relapse risk
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — liver encymes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Alcohol- dependent patients: Detoxified alcohol- dependent patients in an inpatient setting
- Control group: Age- and gender matched healthy controls

SUMMARY:
The aim of this project is to assess which behavioral and neuroimaging alterations associated with reward- based learning predict relapse in alcohol- dependent patients within a follow- up period of 12 months.

The investigators will explore how these alterations interact with clinical and psychosocial factors which can modify the relapse risk. Functional magnetic resonance imaging (fMRI) and positron emission tomography (PET) will be used to identify neurofunctional abnormalities in neurotransmitter systems. The investigators will also provide data for genetic analysis and modeling.

Patients will be detoxified in an inpatient setting and followed for 12 months using the Time-Line Follow- Back Procedure. Clinical assessments, behavioral paradigms of learning and brain imaging will be carried out within at least 4 half- lives after any psychotropic medication.

The investigators will implement and apply functional imaging paradigms assessing Pavlovian-to-instrumental transfer and reversal learning tasks and associate model parameters of learning with alcohol craving, intake and prospective relapse risk.

DETAILED DESCRIPTION:
This project will examine 150 detoxified alcohol-dependent patients and 100 age- and gender matched controls. The main aim of this project is to assess 1) which behavioural and neuroimaging alterations (fMRI) associated with reward-based learning (see Projects 1 & 3) predict relapse within the follow-up period of 6 months, 2) how these interact with clinical and psychosocial factors which can modify the relapse risk, and 3) to provide data for genetic and imaging analyses and modelling. Furthermore, we will explore gender effects on functional imaging parameters of learning. Patients will be detoxified in an inpatient setting and followed for 6 months using the Form 90 and Time-Line Follow-Back Procedure. Clinical assessments, behavioral paradigms of learning, and brain imaging will be carried out within at least 4 half-lives after any psychotropic medication. Subjects will undergo medical management with bimonthly follow-ups and predefined in- and exclusion criteria as described previously. We will implement and apply functional imaging paradigms assessing Pavlovian-to-instrumental transfer and reversal learning as described in Projects 1 and 3. We will associate model parameters of learning with alcohol craving, intake and prospective relapse risk. Independent of these central questions, we will also assess comorbidity, psychosocial and neurobiological disease severity markers to control for specificity of findings.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependence according to DSM-IV
* Minimum of 72 hours of abstinence, maximum of 21 days of abstinence
* Minimum of three years of alcohol dependence
* Low severity of withdrawal symptoms
* Ability to provide fully informed consent and to use self- rating scales

Exclusion Criteria:

* Lifetime history of DSM- IV bipolar or psychotic disorder
* Current threshold DSM-IV diagnosis of any following disorders: current major - depressive disorder, generalized anxiety disorder, PTSD, borderline personality disorder or obsessive- compulsive disorder
* History of substance dependence other than alcohol or nicotine dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Detoxified alcohol- dependent patients and age- and gender matched healthy controls living in Germany
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2012-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
blood oxygenation level dependent (BOLD) response | first assessment time point (alc. dependent pat. up to 21 days after detoxification)
  investigation of neuronal activation of the mesolimbic system in alcohol-dependent patients and healthy controls using 3 Tesla magnetic resonance imaging

SECONDARY OUTCOMES:
Treatment response | 12-month follow-up period beginning after first assessment timepoint
  test the predictive effects of learning parameters and related neuronal correlates for treatment outcome (relapse vs abstinence) in alcohol-dependent patients

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Heinz, Prof MD, Principal Investigator — Charite University, Berlin, Germany; Ulrich S Zimmermann, MD, Principal Investigator — University Hospital Carl Gustav Carus, Dresden, Germany; Andreas Heinz, Prof MD, Study Chair — Charité University, Berlin, Germany; Hans-Ulrich Wittchen, Prof PhD, Study Director — Technische Universität Dresden, Dresden, Germany
Locations (3):
- Germany (3):
  - Technische Universität Dresden, Dresden, Saxony
  - Universitaetsklinikum Carl Gustav Carus at the Technische Universitaet Dresden, Dresden, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin

REFERENCES:
- [Derived] Spitta G, Fliedner LE, Gleich T, Zindler T, Sebold M, Buchert R, Heinz A, Gallinat J, Friedel E. Association between DRD2/ANKK1 TaqIA Allele Status and Striatal Dopamine D2/3 Receptor Availability in Alcohol Use Disorder. J Integr Neurosci. 2022 Oct 28;21(6):171. doi: 10.31083/j.jin2106171. PMID 36424756
- [Derived] Zindler T, Frieling H, Fliedner L, Veer IM, Neyazi A, Awasthi S, Ripke S, Walter H, Friedel E. How alcohol makes the epigenetic clock tick faster and the clock reversing effect of abstinence. Addict Biol. 2022 Sep;27(5):e13198. doi: 10.1111/adb.13198. PMID 36001430
- [Derived] Sebold M, Spitta G, Gleich T, Dembler-Stamm T, Butler O, Zacharias K, Aydin S, Garbusow M, Rapp M, Schubert F, Buchert R, Gallinat J, Heinz A. Stressful life events are associated with striatal dopamine receptor availability in alcohol dependence. J Neural Transm (Vienna). 2019 Sep;126(9):1127-1134. doi: 10.1007/s00702-019-01985-2. Epub 2019 Feb 12. PMID 30747311
- [Derived] Schad DJ, Garbusow M, Friedel E, Sommer C, Sebold M, Hagele C, Bernhardt N, Nebe S, Kuitunen-Paul S, Liu S, Eichmann U, Beck A, Wittchen HU, Walter H, Sterzer P, Zimmermann US, Smolka MN, Schlagenhauf F, Huys QJM, Heinz A, Rapp MA. Neural correlates of instrumental responding in the context of alcohol-related cues index disorder severity and relapse risk. Eur Arch Psychiatry Clin Neurosci. 2019 Apr;269(3):295-308. doi: 10.1007/s00406-017-0860-4. Epub 2018 Jan 8. PMID 29313106
- See also: English study description — http://gepris.dfg.de/gepris/projekt/209290463